CLINICAL TRIAL: NCT00291382
Title: A Multicentre, Stratified, Randomised, Double Blind, Parallel Group Trial to Evaluate Whether a Treatment Strategy Based on Aiming for Total Control Results in Better AHR Than a Treatment Strategy Based on Maintaining Well Control
Brief Title: Airway Hyper-responsiveness Study In Asthma Using Salmeterol/Fluticasone Propionate Combination Product
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: SAM49071
Record Dates: First submitted 2006-02-13; First posted 2006-02-14 (Estimated); Last update posted 2017-05-30 (Actual); Status verified 2017-05

CONDITIONS: Asthma
Keywords: Total asthma control; airway hyper-responsiveness; adult; Asthma
MeSH Terms: conditions — Asthma; Respiratory Hypersensitivity | interventions — Fluticasone-Salmeterol Drug Combination

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: Salmeterol/fluticasone propionate combination

SUMMARY:
This double-blind, stratified, parallel group study is to determine whether aiming for 'Total control' results in better airway hyper-responsiveness than maintaining the treatment level at which 'Well-controlled' asthma was achieved. The primary endpoint is the mean change in PC20 methacholine. Well controlled subjects (as assessed after a 12 week run-in period) will enter a 24 week treatment period during which they will record PEF(Peak Expiratory Flow), symptoms, rescue beta2-agonist use over 24 hours, night time awakenings, asthma exacerbations, emergency visits due to asthma and Adverse Events. At every visit lung function measurements and airway hyper-responsiveness will be measured.

DETAILED DESCRIPTION:
A multi-centre, randomised, double blind, stratified, and parallel group study to evaluate whether a treatment strategy based on aiming for 'Total control' results in better airway hyper-responsiveness than a treatment strategy based on maintaining the treatment level at which 'Well-controlled' asthma was achieved.

ELIGIBILITY:
Inclusion criteria:

* History of asthma of at least 6 months.
* Subjects who have received fluticasone propionate at a dose of 100 mcg bd to 250 mcg bd or equivalent with or without a long acting beta2-agonist for at least 4 weeks before the start of the run-in period, at a constant dose.
* Subjects who are able to understand and complete an electronic diary card.

Exclusion criteria:

* Subjects who have been hospitalized for their asthma within 4 weeks of study entry.
* Subjects who had an acute upper respiratory tract infection within 4 weeks or a lower respiratory tract infection within 4 weeks prior to study entry.
* Subjects who received oral, parental or depot corticosteroids within 4 weeks prior to study entry.
* Subjects who have a known respiratory disorder other than asthma and/or systemic/thoracic abnormalities which influence normal lung function.
* Subjects who have more than 5 pack years.
* Subjects who currently smoke.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Actual)
Dates: Start 2005-11 (Actual); Primary Completion 2007-07 (Actual); Study Completion 2007-07 (Actual)

PRIMARY OUTCOMES:
Mean change in PC20 methacholine (as a measure of airway hyper-responsiveness) following 24 weeks of treatment.

SECONDARY OUTCOMES:
Number of 'Totally-controlled' and Well-controlled patients at the end of the run-in and treatment period according to the GOAL criteria.

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, MD, Study Director — GlaxoSmithKline
Locations (32):
- Belgium (2):
  - GSK Investigational Site, Ghent
  - GSK Investigational Site, Liège
- GSK Investigational Site, Tartu, Estonia
- Finland (2):
  - GSK Investigational Site, Jyväskylä
  - GSK Investigational Site, Tampere
- France (3):
  - GSK Investigational Site, Lille
  - GSK Investigational Site, Montpellier
  - GSK Investigational Site, Poitiers
- Germany (3):
  - GSK Investigational Site, Sinsheim, Baden-Wurttemberg
  - GSK Investigational Site, Bonn, North Rhine-Westphalia
  - GSK Investigational Site, Berlin
- Italy (6):
  - GSK Investigational Site, Foggia, Apulia
  - GSK Investigational Site, Cagliari, Sardinia
  - GSK Investigational Site, Torrette (AN), The Marches
  - GSK Investigational Site, Pisa, Tuscany
  - GSK Investigational Site, Bussolengo (VR), Veneto
  - GSK Investigational Site, Salerno
- GSK Investigational Site, Riga, Latvia
- Netherlands (7):
  - GSK Investigational Site, Breda
  - GSK Investigational Site, Groningen
  - GSK Investigational Site, Harderwijk
  - GSK Investigational Site, Helmond
  - GSK Investigational Site, Hoorn
  - GSK Investigational Site, Nieuwegein
  - GSK Investigational Site, Veldhoven
- Spain (4):
  - GSK Investigational Site, Barcelona
  - GSK Investigational Site, Madrid
  - GSK Investigational Site, Tarrasa, Barcelona
  - GSK Investigational Site, Valencia
- Sweden (3):
  - GSK Investigational Site, Gothenburg
  - GSK Investigational Site, Linköping
  - GSK Investigational Site, Lund